CLINICAL TRIAL: NCT00347945
Title: A Randomized Clinical Trial of Pencil Push-Ups Versus Office Based Vision Therapy For the Treatment of Convergence Insufficiency
Brief Title: Randomized Trial of Treatments for Convergence Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pennsylvania College of Optometry (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HMS2040; 1R21EY13164-1; 1R21EY013164 (NIH)
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2002-01

CONDITIONS: Convergence Insufficiency
Keywords: convergence insufficiency, vision therapy, orthoptics
MeSH Terms: conditions — Ocular Motility Disorders

INTERVENTIONS:
Procedure: Pencil Push-ups
Procedure: Office-based Vision Therapy
Procedure: Placebo Office-based Vision Therapy

SUMMARY:
The Convergence Insufficiency Treatment Trial (CITT) is a multi-center, placebo-controlled, single-masked, clinical trial designed to compare the benefits of two commonly used treatment approaches for patients with convergence insufficiency (CI)

DETAILED DESCRIPTION:
Considerable controversy exists regarding the best treatment for convergence insufficiency (CI), a common condition that often interferes with the ability to perform near work. The two most widely used treatments have significant differences in costs and in practitioner perceived utility. Pencil push-up therapy (PPT) is a simple, low-cost treatment in which patients are prescribed a single procedure to perform at home with only periodic follow-up. Office-based vision therapy (OBVT) is a more comprehensive, time-consuming, complex, and costly treatment in which patients are scheduled for weekly in-office therapy visits and are often prescribed a specific sequence of therapeutic procedures to perform at home. It is important to consider whether either, neither, or both treatments are effective.

The Convergence Insufficiency Treatment Trial (CITT) is a prospective, masked-examiner, multi-center clinical trial in which patients are randomized to one of these two treatment approaches. The primary goal is to answer the following question:

After 12 weeks of treatment, is one therapy more effective than the other in improving CI signs and symptoms? We will test the null hypothesis that there is no difference in the distribution of outcomes between the two populations.

The primary outcome measure will be a classification of each patient as a "success," "improvement," or "failure." This classification will be based on the level of improvement in both the signs (near point of convergence and positive fusional vergence) and symptoms of CI.

Additional questions relate to longer term effects:

1. Are the patients who were classified as "success" or "improvement" at twelve weeks the same at the one-year follow-up for each treatment group?
2. Are there differences in the distributions of changes in near point of convergence, positive fusional vergence, or accommodative amplitudes, between the two treatment groups, at twelve weeks and at one-year of follow up?

ELIGIBILITY:
Inclusion Criteria:

* Age 9-30 years
* Best corrected visual acuity of 20/25 in both eyes at distance and near
* Willingness to wear eyeglasses or contact lenses to correct refractive error, if necessary
* Exophoria at near at least 4 prism diopters greater than at far
* Insufficient positive fusional convergence (i.e., failing Sheard's criterion or minimum normative positive fusional vergence (PFV) of 15 base-out break).
* Receded near point of convergence of > 6 cm break.
* Normal random dot stereopsis using a 500 seconds of arc target.
* CI Symptom Survey score > 16 for subjects in 9-18 year age range and > 21 for subjects in the 19-30 year age range.
* Informed consent and willingness to participate in the study and be randomized

Exclusion Criteria:

* CI previously treated with pencil push-ups (no more than 2 months of treatment within the past year)
* CI previously treated with office-based vision therapy/orthoptics (no more than 2 months of treatment within the past year)
* Amblyopia
* Constant strabismus
* History of strabismus surgery
* Anisometropia >1.50D difference between eyes
* Prior refractive surgery
* Vertical heterophoria greater than 1 
* Systemic diseases known to affect accommodation, vergence, and ocular motility such as: multiple sclerosis, Graves's thyroid disease, myasthenia gravis, diabetes, and Parkinson disease
* Any ocular or systemic medication known to affect accommodation or vergence
* Monocular accommodative amplitude less than 4 D in either eye as measured by the Donder's push-up method
* Manifest or latent nystagmus
* Attention deficit hyperactivity disorder (ADHD) or learning disability diagnosis by parental report
* Household member or sibling already enrolled in the CITT
* Any eye care professional, technician, medical student, or optometry student

Ages: 9 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90
Dates: Start 2000-10; Study Completion 2001-11

PRIMARY OUTCOMES:
The primary outcome measure is the score on the Convergence Insufficiency Symptom Survey

SECONDARY OUTCOMES:
Near Point of Convergence
Positive Fusional Vergence at Near

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Scheiman, OD, Study Chair — Pennsylvania College of Optometry
Locations (7):
- United States (7):
  - Southern California College of Optometry, Fullerton, California
  - State University of New York, College of Optometry, New York, New York
  - The Ohio State University, Optometry Coordinating Center, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Pacific University College of Optometry, Forest Grove, Oregon
  - Eye Institute, Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - University of Houston, College of Optometry, Houston, Texas

REFERENCES:
- [Background] Borsting EJ, Rouse MW, Mitchell GL, Scheiman M, Cotter SA, Cooper J, Kulp MT, London R; Convergence Insufficiency Treatment Trial Group. Validity and reliability of the revised convergence insufficiency symptom survey in children aged 9 to 18 years. Optom Vis Sci. 2003 Dec;80(12):832-8. doi: 10.1097/00006324-200312000-00014. PMID 14688547
- [Background] Gallaway M, Scheiman M, Malhotra K. The effectiveness of pencil pushups treatment for convergence insufficiency: a pilot study. Optom Vis Sci. 2002 Apr;79(4):265-7. doi: 10.1097/00006324-200204000-00013. PMID 11999152
- [Background] Scheiman M, Cooper J, Mitchell GL, de LP, Cotter S, Borsting E, London R, Rouse M. A survey of treatment modalities for convergence insufficiency. Optom Vis Sci. 2002 Mar;79(3):151-7. doi: 10.1097/00006324-200203000-00009. PMID 11913841
- [Result] Scheiman M, Mitchell GL, Cotter S, Cooper J, Kulp M, Rouse M, Borsting E, London R, Wensveen J; Convergence Insufficiency Treatment Trial Study Group. A randomized clinical trial of treatments for convergence insufficiency in children. Arch Ophthalmol. 2005 Jan;123(1):14-24. doi: 10.1001/archopht.123.1.14. PMID 15642806
- [Result] Scheiman M, Mitchell GL, Cotter S, Kulp MT, Cooper J, Rouse M, Borsting E, London R, Wensveen J. A randomized clinical trial of vision therapy/orthoptics versus pencil pushups for the treatment of convergence insufficiency in young adults. Optom Vis Sci. 2005 Jul;82(7):583-95. doi: 10.1097/01.opx.0000171331.36871.2f. PMID 16044063
- [Derived] Scheiman M, Kulp MT, Cotter SA, Lawrenson JG, Wang L, Li T. Interventions for convergence insufficiency: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 2;12(12):CD006768. doi: 10.1002/14651858.CD006768.pub3. PMID 33263359